CLINICAL TRIAL: NCT06761248
Title: Clinical Effectiveness of Fluorescent Starch Nanoparticles Caries Detection Rinse Versus International Caries Detection and Assessment System for Detection of Early Dental Caries in Children: a Diagnostic Accuracy Study
Brief Title: Comparing Fluorescent Starch Nanoparticles Rinse with ICDAS for Early Caries Detection in Children
Acronym: FSNCDR-ICDAS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar kamel salem Eshbair, Doctor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FSN-CDR Vs ICDAS
Record Dates: First submitted 2024-12-27; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Dental Caries; Detection; Fluorescence; Diagnostic Accuracy
Keywords: Fluorescence-Based Caries Detection; Caries Detection Rinse; Early Caries Detection; ICDAS; FSN
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Fluorescent Starch Nanoparticles Rinse for Caries Detection (Experimental): Participants in this arm will undergo diagnostic evaluation using the fluorescent starch nanoparticles caries detection rinse. The rinse contains fluorescent starch nanoparticles that infiltrate porous enamel in active caries lesions. After application, a dental curing light will be used to activate fluorescence, allowing clinicians to identify and differentiate active caries from inactive lesions and other conditions like hypomineralization.
  The performance of the rinse will be compared to the International Caries Detection and Assessment System (ICDAS), which serves as the reference standard for evaluating early dental caries. Data on sensitivity, specificity, and diagnostic accuracy will be collected for analysis.
  Interventions: Device: Fluorescent Starch Nanoparticles Caries Detection Rinse

INTERVENTIONS:
Device: Fluorescent Starch Nanoparticles Caries Detection Rinse — The fluorescent starch nanoparticles caries detection rinse is an innovative diagnostic tool designed to enhance the early detection of active dental caries. It contains proprietary fluorescent starch nanoparticles that infiltrate the porous enamel of active caries lesions. Upon illumination with a standard dental curing light, the nanoparticles fluoresce, allowing clinicians to differentiate active caries from inactive lesions and other enamel conditions. This rinse is evaluated as a non-invasive, highly sensitive, and specific diagnostic device.
  Other Names: LumiKids™ Rinse GreenMark Biomedical

SUMMARY:
The present study aims to evaluate the diagnostic accuracy of fluorescent starch nanoparticles caries detection rinse versus the International Caries Detection and Assessment System (ICDAS) in identifying early dental caries among children from 6 to 11 years old.

DETAILED DESCRIPTION:
Dental caries is a prevalent chronic disease affecting people of all ages globally. It results from the demineralization of tooth enamel and dentin caused by acids produced by bacterial fermentation of dietary sugars in dental plaque. Left untreated, dental caries can progress, leading to pain, infection, and tooth loss. In children, severe caries can interfere with eating, speaking, and learning, while adults may suffer from decreased work performance and lower self-esteem due to poor oral health Early and accurate diagnosis of dental caries is critical for effective management and prevention of disease progression. Detecting caries at an initial stage allows for minimally invasive treatments, such as remineralization therapies, which can arrest or reverse the carious process and prevent the need for extensive restorative procedures. Accurate diagnosis is essential for preserving tooth structure, reducing treatment costs, and improving overall oral health outcomes. Consequently, reliable diagnostic methods are a fundamental aspect of clinical practice, ensuring timely identification and management of caries Traditional caries detection methods, such as visual-tactile examination and radiography, have significant limitations. Visual-tactile examination relies on the clinician's experience and subjective judgment, leading to variability and often missing early caries lesions. Radiographic techniques, useful for detecting interproximal and advanced caries, expose patients to ionizing radiation and may not effectively identify early or non-cavitated lesions. These methods also struggle to detect subsurface demineralization and distinguish between active and inactive lesions, which are critical for effective treatment planning. These limitations highlight the need for more advanced and precise diagnostic tools Fluorescent starch nanoparticles caries detection rinse is an innovative diagnostic tool designed to enhance the detection of active dental caries. It utilizes proprietary fluorescent starch nanoparticles that infiltrate the porous enamel of active lesions. When illuminated with a dental curing light, these nanoparticles fluoresce, allowing clinicians to distinguish active caries from inactive lesions and other conditions like hypomineralization. This rinse provides high sensitivity, specificity, and diagnostic accuracy, addressing limitations in conventional visual-tactile and radiographic methods. LumiCare is an approach to improving early caries diagnosis, aligning with minimally invasive dentistry principles

ELIGIBILITY:
Inclusion Criteria:

* Children with active initial caries.
* At least two teeth with active caries (ICDAS 1 or 2) and two teeth with inactive caries.

Exclusion Criteria:

* Teeth with hypoplasia, fractures, or conditions like dentinogenesis imperfecta.
* Children with fixed orthodontic appliances.
* Participants whose guardians refuse consent.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | through study completion, an average of 1 year
  Measured using sensitivity, specificity, positive predictive value, and negative predictive value.

CONTACTS AND LOCATIONS:
Overall Officials: Associate Prof. Dr. Mariam Mohsen aly, Ph.D., Study Director — Cairo University; Dr. Reem Mohamed Fouad Wahby, Ph.D., Study Chair — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Giza Governorate, Egypt

REFERENCES:
- [Background] Deeks JJ, Altman DG. Diagnostic tests 4: likelihood ratios. BMJ. 2004 Jul 17;329(7458):168-9. doi: 10.1136/bmj.329.7458.168. No abstract available. PMID 15258077
- [Background] Amaechi BT, Phillips TS, Perozo BI, Kataoka Y, Movaghari Pour F, Farah R, Obiefuna AC, Farokhi MR. Evaluation of a novel caries detecting oral rinse. BDJ Open. 2023 Mar 20;9(1):12. doi: 10.1038/s41405-023-00134-y. PMID 36941251